CLINICAL TRIAL: NCT04701216
Title: A Phase 1 Open-Label Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of SHR8735 in Healthy Chinese and Caucasian Subjects
Brief Title: A Trial of SHR8735 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR8735-I-113
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: SHR8735 cohort 1 (Experimental): The subjects will receive a multiple dose of SHR8735 (low dose).
  Interventions: Drug: SHR8735
- Experimental: SHR8735 cohort 2 (Experimental): The subjects will receive a single dose of SHR8735 (medium dose).
  Interventions: Drug: SHR8735
- Experimental: SHR8735 cohort 3 (Experimental): The subjects will receive a single dose of SHR8735 (high dose).
  Interventions: Drug: SHR8735

INTERVENTIONS:
Drug: SHR8735 — SHR8735 is an thrombopoietin receptor agonist to promote platelet production.

SUMMARY:
This is a phase 1 open-label study.

DETAILED DESCRIPTION:
This is a phase 1 open-label study. The objective of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of oral administered SHR8735 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial, and provides written informed consent.
* Be able to comply with all the requirements and able to complete the study.
* Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
* No clinically significant abnormalities in medical history, general physical examination, vital signs, and laboratory tests.
* Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods and have no plan to have a child from signing the consent form to 16 weeks after IP administration.

Exclusion Criteria:

* Receipt of any other investigational drugs or medical devices within 3 months prior to screening (according to the date of signed consent form).
* History of illicit or prescription drug abuse or addiction within one year of screening, or positive urine drug screen at screening and Day-1. The urine drug screen may be repeated at the discretion of the investigator and the reason for repeat needs to be documented clearly (e.g., suspicion of false positive due to diet).
* Severe, active psychiatric conditions that require ongoing treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 28 days)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 15 days)
  Area under the concentration-time curve from time 0 to last time point after SHR8735 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 15 days)
  Area under the concentration-time curve from time 0 to infinity after SHR8735 administration
Pharmacokinetics-Tmax | Up to 15 days
  Time to Cmax of SHR8735
Pharmacokinetics-Cmax | Up to 15 days
  Maximum observed concentration of SHR8735
Pharmacokinetics-CL/F | Up to 15 days
  Apparent clearance of SHR8735
Pharmacokinetics-Vz/F | Up to 15 days
  Apparent volume of distribution during terminal phase of SHR8735
Pharmacokinetics-t1/2 | Up to 15 days
  Terminal elimination half-life of SHR8735
Change from baseline to end of treatment for platelet count | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana Sun, Dr, Principal Investigator — Study Principal Investigator
Locations (1):
- Linear Clinical research, Perth, Western Australia, Australia